CLINICAL TRIAL: NCT00277550
Title: A Randomized, Double-blind, Placebo-controlled Evaluation of the Effects of Tegaserod (6 mg b.i.d) on Whole Gut Transit Time in Patients With Chronic Idiopathic Constipation and Dyspepsia
Brief Title: The Effects of Tegaserod vs. Placebo on Whole Gut Transit Time in Patients With Chronic Constipation and Dyspepsia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919EUS42
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Constipation and Dyspepsia
Keywords: Constipation, Tegaserod, Dyspepsia
MeSH Terms: conditions — Constipation; Dyspepsia | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod and Placebo

SUMMARY:
To demonstrate the effects of tegaserod on gastrointestinal scintigraphic orocecal transit in female patients with CC and upper GI symptoms of dyspepsia

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 to 64 years of age
* Patients must present with two or more of the following criteria for chronic constipation for at least 12 weeks prior to entering the study:

  1. Less than 3 bowel movements per week
  2. Hard or lumpy stools
  3. Straining during bowel movements
  4. Feeling of incomplete evacuation
* Patients must report overlapping symptoms consistent with dyspepsia, such as mid-upper abdominal discomfort characterized by early satiety, post-meal fullness and bloating

Exclusion Criteria:

* Patients with a recent history of, or current frequency of diarrhea occuring more than once per month off of laxatives
* Clinically significant diagnosis of pelvic outlet obstruction or pelvic floor dyssenergia as determined by the study physicians
* Patients with constipation secondary to medication use as determined by the study physician
* Patients with clinically significant abnormal TSH levels at screening
* Patients that have heartburn or abdominal pain as their predominant GI symptom
* Evidence of cathartic colon or a history of laxative abuse

  * Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To determine the effect of one week of tegaserod on the passage of content through the gut by radiological procedures.

SECONDARY OUTCOMES:
To evaluate the PD effects of tegaserod on upper & lower GI transit
To evaluate global well-being & upper and lower GI symptoms in daily assessment of bowel habits and weekly global and individual symptom assessments

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Talley, MD, Principal Investigator — Mayo Clinic; Michael Crowell, PhD, Principal Investigator — Mayo Clinic